CLINICAL TRIAL: NCT05924724
Title: Prospective, Randomized Pilot Study to Improve the Treatment Satisfaction and Treatment Adherence of Diabetic Women Through the Use of Flash Glucose Monitoring Systems
Brief Title: Treatment Satisfaction and Treatment Adherence of Diabetic Women Through the Use of FGM
Acronym: Flash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Flash
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes; Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes; GDM; FGM; Flash Glucose Monitoring; SMBG; self monitoring of blood glucose
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage Flash-Glucose Monitoring FGM (Experimental): Participants in this arm will transition from routine care using SMBG to using FGM after one week. They will receive training on how to use the FGM device. The FGM will be used continuously from that point until delivery, throughout the entire pregnancy.
  Interventions: Device: Flash Glucose Monitoring
- Usage Self-Monitoring Blood Glucose SMBG (No Intervention): Participants in this arm will remain in the routine care using SMBG. They will use it continuously from diagnosis until delivery, throughout the entire pregnancy.

INTERVENTIONS:
Device: Flash Glucose Monitoring — The FGM is a non-invasive device typically worn on the upper arm, designed to continuously measure blood glucose levels without the need for fingerstick capillary measurements.
  Arms: Usage Flash-Glucose Monitoring FGM

SUMMARY:
The incidence of gestational diabetes mellitus (GDM), a glucose tolerance disorder during pregnancy, is increasing. In Germany, it reached 8.58 % in 2019. Standardized treatment has reduced complications for mother and child. Blood self-measurement is currently used to monitor glucose levels, but it is burdensome and disliked by patients. Flash Glucose Monitoring (FGM) was approved in 2017, but its routine use lacks sufficient data. This pilot project aims to study the impact of FGM on patient satisfaction and adherence to therapy. The hypothesis is that FGM will improve patient experience and increase therapy adherence. The study will include 100 GDM-diagnosed women who will be randomly assigned to FGM or SMBG treatment. The primary endpoint is treatment satisfaction and adherence, measured through step count, physical activity, food error count, and weight gain. The project aims to provide data for patient-centered decision-making on glucose monitoring systems, following the principles of the Association of Diabetes Counseling and Training Professions in Germany (VDBD).

DETAILED DESCRIPTION:
The incidence of gestational diabetes mellitus (GDM), defined as a glucose tolerance disorder diagnosed for the first time during pregnancy, is steadily increasing, reaching 8.58 % in Germany in 2019, according to figures from the Institute for Quality Assurance and Transparency in Health Care (IQTIG). Standardized guideline-compliant treatment has significantly reduced the rate of perinatal complications for both mother and child. A central component of management is the adjustment of blood glucose levels to the specified target values. To date, patients' glucose levels have been determined by blood self-measurement (SMBG) in accordance with guidelines. The diagnosis of GDM and the subsequent management is perceived by the patients as an enormous burden, especially because of the self-measurement, which is perceived as time-consuming, painful and stigmatizing. Since 2017, the Flash Glucose Monitoring (FGM) has been approved for use in the care of pregnant diabetic women. Its use by gestational diabetics is critically discussed. To date, there is a lack of systematically collected data on the use of FGM in the care of GDM patients that would justify its routine use.

The aim of the pilot project planned here is to investigate the influence of FGM on patient satisfaction and adherence to therapy. The investigators hypothesize that the use of the FGM relieves the affected women decisively and mediated by biofeedback leads to more therapy adherence. These data will be used to plan a multicenter study.

At the Competence Center for Diabetes and Pregnancy of the University Hospital Jena, 100 women diagnosed with GDM will be included in a randomized controlled trial and will be treated with either FGM (n = 50) or SMBG (n = 50) and followed up according to the guidelines.

The primary endpoint is the assessment of treatment satisfaction and adherence using the following measures: step count, physical activity (IPAQ), food error count and weight gain.

In order to meet the principle "In the sense of a patient-centered individual therapy, the affected persons should be involved in the decision for or against a glucose monitoring system" of the Association of Diabetes Counseling and Training Professions in Germany (VDBD), the aim of our project is to create a data basis for this.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age above 18 years
* single cephalic pregnancy
* newly diagnosed gestational diabetes mellitus
* 24+0 - 30+0 weeks of gestation

Exclusion Criteria:

* severe pregnancy complications
* severe fetal malformations
* rejection of FGM device by health care provider
* existing diabetes mellitus (type 1 or type 2)
* glucose metabolism affecting diseases
* bariatric surgeries in the past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction | The questionnaire will be filled by the participant during 33 to 35 weeks of gestation.
  The treatment satisfaction is anticipated to be evaluated using the Diabetes Treatment Satisfaction Questionnaire change (DTSQc) with minimal value of -18 and maximal value of 18, with higher values indicating more satisfaction.

SECONDARY OUTCOMES:
Step Count per Day | daily starting at 24 weeks of gestation until delivery
  Step count will be documented by the participant and will be evaluated as progression. It is advised, that patients diagnosed with diabetes aim to increase their step count.
Activity in the last 7 days | every two weeks starting at 24 weeks of gestation until delivery
  The activity is evaluated using the international physical activity questionnaire (IPAQ). The Score provides the metabolic equivalent of task (MET)-minutes per week in total, with a minimum of 0 and a maximum of 100.000 MET-min/week. Higher score indicate higher activity.

CONTACTS AND LOCATIONS:
Overall Officials: Friederike Weschenfelder, Dr., Principal Investigator — University Hospital Jena, Department of Obstetrics
Locations (1):
- Universitätsklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No